CLINICAL TRIAL: NCT00886379
Title: Blue Sky Study: Impact of Milk and Vitamin D for Child Growth and Health
Acronym: BSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Janet Rich-Edwards, Direct of Developmental Epidemiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSS-103306
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Vitamin d Deficiency
Keywords: vitamin d; children; Mongolia
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Milk Substitutes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): Mongolian milk without D
  Interventions: Dietary Supplement: Mongolian milk without vitamin D
- 2 (Experimental): Mongolian milk with vitamin D
  Interventions: Dietary Supplement: Mongolian milk with vitamin D
- 3 (Experimental): Ultra High Temperature (UHT) milk
  Interventions: Dietary Supplement: UHT milk
- 4 (Experimental): Milk Substitute
  Interventions: Dietary Supplement: Milk Substitute
- 5 (Experimental): Seasonal D
  Interventions: Dietary Supplement: Seasonal D supplement
- 6 (Experimental): Daily D
  Interventions: Dietary Supplement: Daily D supplement

INTERVENTIONS:
Dietary Supplement: Mongolian milk without vitamin D — 710ml per day for 49 days
  Other Names: Guum milk
  Arms: 1
Dietary Supplement: Mongolian milk with vitamin D — 710ml per day for 49 days. A total of 13,700 IU of vitamin D over the intervention period.
  Other Names: Guum milk
  Arms: 2
Dietary Supplement: UHT milk — 710ml per day for 49 days. A total of 13,700 IU of vitamin D over the intervention period.
  Other Names: Gossner milk
  Arms: 3
Dietary Supplement: Milk Substitute — 710ml per day for 49 days. A total of 13,700 IU of vitamin D over the intervention period.
  Other Names: Mead Johnson
  Arms: 4
Dietary Supplement: Seasonal D supplement — Deliver dosage of 13,700 IU vitamin D over 7 days
  Other Names: Tish Con
  Arms: 5
Dietary Supplement: Daily D supplement — Deliver dosage of 13,700 IU vitamin D in vitamin capsules over 49 days.
  Other Names: Tish Con
  Arms: 6

SUMMARY:
This intervention study will address the impact of vitamin D fortified milk and vitamin D supplements on the growth, levels of vitamin D, insulin-like growth factor 1, growth hormone, academic attention, respiratory infections, asthma, and flexural dermatitis (a proxy for eczema) of Mongolian children.

ELIGIBILITY:
Inclusion Criteria:

* Children in 3rd and 4th grade from selected Mongolian schools.
* School selection will consider:

  * socioeconomic position;
  * geographic location;
  * school size;
  * current lunch or supplementation program; and
  * the interest and willingness to participate of the school's administration and faculty.

Exclusion Criteria:

* Allergy to milk or wheat products.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 597 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rich-Edwards, Sc.D., Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Background] Rich-Edwards JW, Ganmaa D, Pollak MN, Nakamoto EK, Kleinman K, Tserendolgor U, Willett WC, Frazier AL. Milk consumption and the prepubertal somatotropic axis. Nutr J. 2007 Sep 27;6:28. doi: 10.1186/1475-2891-6-28. PMID 17900364
- [Derived] Rich-Edwards JW, Ganmaa D, Kleinman K, Sumberzul N, Holick MF, Lkhagvasuren T, Dulguun B, Burke A, Frazier AL. Randomized trial of fortified milk and supplements to raise 25-hydroxyvitamin D concentrations in schoolchildren in Mongolia. Am J Clin Nutr. 2011 Aug;94(2):578-84. doi: 10.3945/ajcn.110.008771. Epub 2011 Jun 22. PMID 21697075

RESULTS

PARTICIPANT FLOW:
Groups:
- Unfortified Mongolian Milk: Mongolian milk without vitamin D: 710ml per day for 49 days
- Fortified Mongolian Milk: Mongolian milk with vitamin D: 710ml per day for 49 days. A total of 13,700 IU of vitamin D over the intervention period.
- Fortified UHT Milk: UHT milk: 710ml per day for 49 days. A total of 13,700 IU of vitamin D over the intervention period.
- Daily Vitamin D Supplements: Daily D supplement: Deliver dosage of 13,700 IU vitamin D in vitamin capsules over 49 days.
- Seasonal Vitamin D Supplements: Seasonal D supplement: Deliver dosage of 13,700 IU vitamin D over 7 days
Period: Overall Study
Arm/Group | Unfortified Mongolian Milk | Fortified Mongolian Milk | Fortified UHT Milk | Daily Vitamin D Supplements | Seasonal Vitamin D Supplements
Started | 104 | 143 | 143 | 112 | 95
Completed | 101 | 140 | 137 | 109 | 92
Not Completed | 3 | 3 | 6 | 3 | 3
Not completed — Transferred Schools | 0 | 0 | 2 | 1 | 1
Not completed — Final blood draw not obtained | 3 | 3 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Unfortified Mongolain Milk: Mongolian milk without vitamin D: 710ml per day for 49 days
- Total: Total of all reporting groups
Arm/Group | Unfortified Mongolain Milk | Fortified Mongolian Milk | Fortified UHT Milk | Daily Vitamin D Supplements | Seasonal Vitamin D Supplements | Total
Number analyzed (Participants) | 101 | 140 | 137 | 109 | 92 | 579
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 101 | 140 | 137 | 109 | 92 | 579
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 65 | 69 | 45 | 41 | 271
  Male | 50 | 75 | 68 | 64 | 51 | 308

OUTCOME MEASURES:

1. Primary Outcome: Serum 25-hydroxyvitamin D Concentrations in Schoolchildren
Description: Baseline and Follow-up 25(OH)D3 by liquid chromatography-tandem mass spectrometry
Time Frame: Blood was analyzed at day 0 and day 49
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Unfortified Mongolain Milk | Fortified Mongolian Milk | Fortified UHT Milk | Daily Vitamin D Supplements | Seasonal Vitamin D Supplements
Number analyzed (Participants) | 101 | 140 | 137 | 109 | 92
ng/ml
  Blood concentration on Day 0 | 8 (4) | 8 (4) | 10 (5) | 7 (3) | 8 (4)
  Blood concentration on Day 49 | 8 (4) | 20 (6) | 29 (10) | 21 (6) | 12 (4)

ADVERSE EVENTS:
Arm/Group | Unfortified Mongolain Milk | Fortified Mongolian Milk | Fortified UHT Milk | Daily Vitamin D Supplements | Seasonal Vitamin D Supplements
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/140 | 0/137 | 0/109 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/140 | 0/137 | 0/109 | 0/92
Other Adverse Events (participants affected / at risk) | 0/101 | 0/140 | 0/137 | 0/109 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes